CLINICAL TRIAL: NCT07146451
Title: 6-year Follow-up of Children Born to Mothers Exposed to Nifedipine vs Placebo After Preterm Prelabor Rupture of Membranes at 22 to 33 Weeks of Gestation
Brief Title: 6-year Outcomes in Children After Nifedipine vs Placebo for Preterm Prelabor Rupture of Membranes at 22-33 Weeks
Acronym: TOCOKIDS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230846
Record Dates: First submitted 2025-07-16; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Children Born to Mothers Enrolled in the TOCOPROM Trial
Keywords: Prematurity; Nifedipine; Psychological assessment; Neurodevelopment; School age; Preterm prelabor rupture of membranes
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nifedipine: Exposure during pregnancy to Oral Nifedipine 20 mg LP (between 22 to 33 weeks of gestation): Loading dose at T0 and T0.5 (i.e. 30 min), total=2x20 mg Maintenance dose:
  Oral Nifedipine 20 mg LP at T3, then 1 pill every 8 hours for 48 hours (i.e. T11, T19, T27, T35 and T43, total=6x20 mg)
  Interventions: Other: Self-administered parental questionnaire
- Placebo: Exposure during pregnancy to oral placebo of nifedipine (between 22 to 33 weeks of gestation) at T0, T0.5, T3, T11, T19, T27, T35 and T43
  Interventions: Other: A short psychological assessment performed online

INTERVENTIONS:
Other: Self-administered parental questionnaire — A self-administered parental questionnaire, completed online or on paper, to assess different dimension of neurodevelopment
  Groups: Nifedipine
Other: A short psychological assessment performed online — NEMI-3: an intelligence test administered by a psychologist measuring a fluid and crystallised intelligence. The test consists of 117 spoken and visual questions, for a total administration time of 45 min. Results are expressed in the form of standard indices (mean 100, standard deviation 15) that facilitate comparisons with the results obtained on other intelligence scales.
  Results will be classified as normal, mild delay (between 1 and <2 standard deviation [SD] below the mean) or severe delay (≥2 SD).
  Groups: Placebo

SUMMARY:
The purpose of this study is to evaluate the neurodevelopment at age 6 of children born to women with preterm prelabor rupture of membranes at 22 to 33 weeks of gestation, after antenatal exposure to nifedipine vs placebo.

DETAILED DESCRIPTION:
Preterm prelabor rupture of membranes (PPROM) complicates 3% of pregnancies and accounts for one-third of preterm births. It is a leading cause of neonatal mortality and morbidity and increases the risk of maternal infectious morbidity. In cases of early PPROM (22 to 33 completed weeks' gestation), expectant management is recommended in the absence of labor, chorioamnionitis or fetal distress. Antenatal steroids and antibiotics administration are recommended by international guidelines. However, there is no recommendation regarding tocolysis administration in the setting of PPROM. In theory, reducing uterine contractility should delay delivery and reduce the risks of prematurity and neonatal adverse consequences. Likewise, a prolongation of gestation may allow administering a corticosteroids complete course that is associated with a two-fold reduction of morbidity and mortality. However, tocolysis may prolong fetal exposure to inflammation and be associated with higher risk of materno-fetal infection, potentially associated with neonatal death or long-term sequelae, including cerebral palsy.

The investigators implemented the TOCOPROM randomized clinical trial to assess whether short-term (48 hr) tocolysis reduces perinatal morti-morbidity in cases of PPROM at 22-33 weeks. However, both short- and long-term outcomes should be taken into account to define the optimal treatment strategy. There are currently no data allowing to evaluate the impact of a short course of nifedipine versus placebo on neurodevelopmental outcomes in school-aged children born after PPROM. Therefore, following-up children born to mothers enrolled in the TOCOPROM trial, through a new study, the TOCOKIDS cohort, is a unique and timely opportunity to advance scientific knowledge and adapt clinical practices in France and worldwide.

The assessment at 6 years of age will consist in:

* A self-administered parental questionnaire, completed online or on paper
* Data collected from the health book, in particular the 6-year consultation
* A short psychological assessment (45 minutes), performed remotely by a psychologist through video conference.

ELIGIBILITY:
Inclusion Criteria:

* All children born to mothers enrolled in the TOCOPROM trial who consented to participate in the 2-year follow-up and who agreed to be contacted for the 6-year follow-up
* Alive at 6 years
* Internet access, including access to a good-quality video-conference system (only for the psychological evaluation)
* Non opposition of the holders of the exercise of parental authority

Exclusion Criteria:

* Major malformations and/or chromosomal aberrations evidenced after birth
* Impossibility to contact the family
* Opposition to participate in the follow-up

Ages: 6 Years to 78 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born to women enrolled in the TOCOPROM trial reaching the age of 6 years
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2033-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Cerebral palsy at 6 years of age. | Up to 6 months after inclusion.
  Cerebral palsy assessed using the Gross Motor Function Classification System (GMFCS), a five-level classification based on the child's current gross motor abilities, limitations in gross motor function, and need for assistive technology and wheeled mobility.
  Severe/moderate cerebral palsy (GMFCS≥2). Mild cerebral palsy (GMFCS-1).
Developmental Coordination Disorder at 6 years of age. | Up to 6 months after inclusion.
  Measured using the Developmental Coordination Disorder Questionnaire - European French (DCDQ-FE), a brief parent questionnaire (15 items) designed to screen for gross and fine motor skills and coordination disorders in children, aged 5 to 15 years.
  Total score=15-56: indication of a risk of DCD or suspected of a risk of DCD. Total score=57-75: probably no DCD.
Language at 6 years of age | Up to 6 months after inclusion.
  Language assessed using the verbal communication subscale (4 items) of the 5-15R scale, covering comprehension, expressive language skills and verbal communication, with an extra question on the impact of language and communication difficulties on daily activities.
  Mean (SD). Reference to cut-off scores in relation to the 90 and 98 percentiles (%).
Behavior at 6 years of age. | Up to 6 months after inclusion.
  Behavior assessed using the Strengths and Difficulties Questionnaire (SDQ), a brief behavioral screening questionnaire (25 items), designed to screen for symptoms of hyperactivity inattention, emotional, conduct, and peer problems among 2-17 year olds.
  Mean (SD). Abnormal: >90th percentile. Mildly abnormal: 80-90 percentile.
Executive functions at 6 years of age. | Up to 6 months after inclusion.
  Executive functions measured using the Childhood Executive Functioning Inventory (CHEXI), a rating instrument (24 items) for parents that was developed for measuring executive functioning in children age 4-12. It includes four different subscales tapping working memory, planning, regulation and inhibition, combined into two global scales: working memory (working memory and planning subscales) and inhibition (inhibition and regulation subscales).
  Normative data are not yet available. Abnormality will be defined considering a cut-off or deviation compared to the mean score, depending on the literature.

SECONDARY OUTCOMES:
Vital status at 6 years of age. | Up to 6 months after inclusion.
  Whether the child is alive or not at years of age.
Neurodevelopmental impairment. | Up to 6 months after inclusion.
  Moderate-to-severe impairment (severe/moderate cerebral palsy, and/or abnormal SDQ score, and/or NEMI-3 ≥2 SD below the mean, and/or blindness, and/or deafness), mild impairment (mildly abnormal scores or mild impairment) vs no neurodevelopmental impairment.
Survival without any neurodevelopmental impairment at 6 years of age. | Up to 6 months after inclusion.
  Survival without any neurodevelopmental impairment (as defined in the primary endpoint, and then including also cognitive impairment).
Survival without moderate-to-severe neurodevelopmental impairment at 6 years of age. | Up to 6 months after inclusion.
  Survival without moderate-to-severe neurodevelopmental impairment (i.e. severe/moderate cerebral palsy, and/or abnormal SDQ score, and/or NEMI-3 ≥2 SD below the mean, and/or blindness, and/or deafness).
Growth at 6 years of age. | Up to 6 months after inclusion.
  Height compulsory examination in the sixth year, reported in the health book.
Growth at 6 years of age | Up to 6 months after inclusion
  Weight. Compulsory examination in the sixth year, reported in the health book
Health at 6 years of age. | Up to 6 months after inclusion.
  Arterial pressure. Compulsory examination in the sixth year, reported in the health book.
Health at 6 years of age | Up to 6 months after inclusion
  chronic diseases, compulsory examination in the sixth year, reported in the health book
Health at 6 years of age | Up to 6 months after inclusion
  oral health. Compulsory examination in the sixth year, reported in the health book
Vision at 6 years of age. | Up to 6 months after inclusion.
  Visual acuity, any vision problem mentioned. Compulsory examination in the sixth year, reported in the health book.
Hearing at 6 years of age. | Up to 6 months after inclusion.
  Hearing test. Compulsory examination in the sixth year, reported in the health book.
Development at 6 years of age. | Up to 6 months after inclusion.
  Data reported in the health book during the compulsory examination in the sixth year.
Language at 6 years of age. | Up to 6 months after inclusion.
  Language test. Compulsory examination in the sixth year, reported in the health book.
Behaviour at 6 years of age. | Up to 6 months after inclusion.
  Data reported in the health book during the compulsory examination in the sixth year.
Cognition at 6 years of age. | Up to 6 months after inclusion.
  NEMI-3: an intelligence test administered by a psychologist measuring a fluid and crystallised intelligence. The test consists of 117 spoken and visual questions, for a total administration time of 45 min. Results are expressed in the form of standard indices (mean 100, standard deviation 15) that facilitate comparisons with the results obtained on other intelligence scales.
  Results will be classified as normal, mild delay (between 1 and <2 standard deviation [SD] below the mean) or severe delay (≥2 SD).
Feasibility of performing an online psychological evaluation. | Up to 6 months after inclusion.
  Acceptability E-Scale (adapted - 3 items), participation and completion rates, technical difficulties.
Parent-reported health and development. | Up to 6 months after inclusion.
  Self-reported. Perceived health and development of the child, parental concerns about health and development, and professional diagnoses of health conditions (e.g., asthma, respiratory problems, etc.).
Parent-reported Health-Related Quality of Life. | Up to 6 months after inclusion.
  PedsQL Short Form - 15 items. All items will be added up and linearly transformed on a scale between 0 and 100, a higher score indicating a better HRQoL. Physical and psychosocial functioning will be further assessed using the corresponding subscales. Poor HRQoL, physical or psychosocial functioning will be defined using thresholds compatible with a severe health condition.
Parent-reported school difficulties | Up to 6 months after inclusion
  Ad-hoc questions
Maternal self-perceived health | Up to 6 months after inclusion
  Minimum European Health Module - 1 item
Maternal mental health | Up to 6 months after inclusion
  PHQ-4 (anxiety and depression) - 4 items
Maternal well-being | Up to 6 months after inclusion
  WHO-5 Well-Being Index - 5 items
Maternal quality of life | Up to 6 months after inclusion
  WHOQOL bref FR - 1 item

CONTACTS AND LOCATIONS:
Overall Officials: Gilles KAYEM, MD,PhD, Principal Investigator — Université Paris Cité and Université Sorbonne Paris Nord, Paris, France. DHU Risks in Pregnancy, Paris Descartes University, Trousseau University Hospital; Elsa LORTHE, RM,PhD, Study Director — Université Paris Cité and Université Sorbonne Paris Nord, Paris, France.
Locations (1):
- Trousseau University Hospital, Paris, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Houtzager BA, Hogendoorn SM, Papatsonis DN, Samsom JF, van Geijn HP, Bleker OP, van Wassenaer AG. Long-term follow up of children exposed in utero to nifedipine or ritodrine for the management of preterm labour. BJOG. 2006 Mar;113(3):324-31. doi: 10.1111/j.1471-0528.2006.00851.x. PMID 16487205
- [Background] Van De Water M, Kessel ET, De Kleine MJ, Oei SG. Tocolytic effectiveness of nifedipine versus ritodrine and follow-up of newborns: a randomised controlled trial. Acta Obstet Gynecol Scand. 2008;87(3):340-5. doi: 10.1080/00016340801913189. PMID 18307075
- [Background] van Vliet E, Seinen L, Roos C, Schuit E, Scheepers H, Bloemenkamp K, Duvekot JJ, van Eyck J, Kok JH, Lotgering FK, van Baar A, van Wassenaer-Leemhuis AG, Franssen MT, Porath MM, van der Post J, Franx A, Mol B, Oudijk MA. Maintenance tocolysis with nifedipine in threatened preterm labour: 2-year follow up of the offspring in the APOSTEL II trial. BJOG. 2016 Jun;123(7):1107-14. doi: 10.1111/1471-0528.13586. Epub 2015 Aug 27. PMID 26330379
- [Background] van Winden T, Klumper J, Kleinrouweler CE, Tichelaar MA, Naaktgeboren CA, Nijman TA, van Baar AL, van Wassenaer-Leemhuis AG, Roseboom TJ, Van't Hooft J, Roos C, Mol BW, Pajkrt E, Oudijk MA. Effects of tocolysis with nifedipine or atosiban on child outcome: follow-up of the APOSTEL III trial. BJOG. 2020 Aug;127(9):1129-1137. doi: 10.1111/1471-0528.16186. Epub 2020 Mar 29. PMID 32124520
- [Background] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046
- [Background] Lorthe E, Kayem G; TOCOPROM Study Group and the GROG (Groupe de Recherche en Obstetrique et Gynecologie). Tocolysis in the management of preterm prelabor rupture of membranes at 22-33 weeks of gestation: study protocol for a multicenter, double-blind, randomized controlled trial comparing nifedipine with placebo (TOCOPROM). BMC Pregnancy Childbirth. 2021 Sep 8;21(1):614. doi: 10.1186/s12884-021-04047-2. PMID 34496799